CLINICAL TRIAL: NCT02827201
Title: Phase II Randomised Multicenter Trial Evaluating a Sequential Treatment With Nab-paclitaxel+Gemcitabine /FOLFIRI.3 vs Nab-paclitaxel + Gemcitabine in First Line Metastatic Pancreatic Cancer
Brief Title: FIrst Line Treatment of Metastatic Pancreatic Cancer: Sequential Nab-paclitaxel + Gemcitabine/FOLFIRI.3 VS Nab-paclitaxel + Gemcitabine
Acronym: FIRGEMAX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Collaborators: UNICANCER (Other); GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRODIGE 37
Record Dates: First submitted 2015-11-26; First posted 2016-07-11 (Estimated); Results first posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nab-paclitaxel + gemcitabine/FOLFIRI.3 (Experimental): Alternance of :
  * 2 months with nab-paclitaxel (125 g/m² - 30 min in IV) + gemcitabine (1000 mg/m², 30 min in IV, 3 injections follow by 1 week free)
  * follow by 2 months with FOLFIRI.3 (irinotecan: 90 mg/m² at D1, acid folinic 400 mg/m², 5Fu continus: 2000 mg/m² IV 46 hours, and irinotecan at D3, 90 mg/m²) This alternance continus until progression
  Interventions: Drug: FOLFIRI.3; Drug: nab-paclitaxel+ gemcitabine
- nab-paclitaxel + gemcitabine (Active Comparator): nab-paclitaxel (125 g/m² - 30 min in IV) + gemcitabine (1000 mg/m² - 30 min in IV) 3 injections follow by 1 week free, until progression
  Interventions: Drug: nab-paclitaxel+ gemcitabine

INTERVENTIONS:
Drug: FOLFIRI.3 — For each cycle : 1 week out of 2 - injection at Day1, J15 Irinotécan 90 mg/m² at day1 in perfusion over 60 min in Y of folinic acid Folinic Acid 400 mg/m² (or 200 mg/m² Elvorine) at Day 1 in perfusion over 2 hours 5FU continu 2000 mg/m² during 46 hours Irinotécan at 90 mg/m² in perfusion over 60 mn at Day 3 (when 5FU perfusion is over)
  Arms: nab-paclitaxel + gemcitabine/FOLFIRI.3
Drug: nab-paclitaxel+ gemcitabine — For each cycle : 3 weeks out of 4 - injection at Day 1, 8 and 15 Nab-paclitaxel : 125 mg/m² of nab-paclitaxel in perfusion over 30 mn. Gemcitabine 1000 mg/m² in perfusion over 30 mn immediately after Nab paclitaxel administration is over.

SUMMARY:
The main objective of this trial is to evaluate every 2 months alternating nab-paclitaxel/gemcitabine and FOLFIRI.3 versus nab-paclitaxel + gemcitabine, regarding the progression of disease at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of pancreatic adenocarcinoma
* Distant metastatic disease
* Scan (or MRI if scanner contraindicated) completed within 3 weeks of the start of treatment
* At least one lesion measurable by RECIST v1.1 criteria
* Life expectancy> 3 months
* No previous chemotherapy (adjuvant chemotherapy with gemcitabine authorised if administered more than 6 months prior to inclusion)
* No previous radiotherapy (unless at least one measurable target lesion outside the irradiation zone)
* Pain must be monitored before inclusion
* 18 years < age < 75
* Performance status: WHO < 2
* ANC ≥ 1500/mm3, platelets ≥ 100 000/mm3, haemoglobin ≥ 9 g/dL
* ASAT (SGOT), ALAT (SGPT) ≤ 2.5 x ULN or ≤ 5 x ULN if liver metastases found
* Bilirubin ≤ 1.5 x ULN (patients drained by retrograde technique are includable), creatinine < 120 μmol/L, or MDRD creatinine clearance > 60 mL/min
* Women of childbearing age must have a negative pregnancy test (β HCG) before starting treatment
* Women of childbearing age as well as men (who have sexual intercourse with women of childbearing age) must agree to use effective contraception without interruption for the duration of treatment and 6 months after the administration of the last treatment dose
* Patient affiliated to the social security scheme
* Patient information and signature of informed consent

Exclusion Criteria:

* - Other types of pancreatic tumours, especially endocrine or acinar cell tumours
* Ampulloma
* Presence of meningeal or cerebral metastases, bone metastases
* Gilbert's syndrome
* Presence of neuropathy> grade 1 according to NCIC-CTC 4.0
* Contraindications specific to the studied treatments
* History of chronic diarrhoea or inflammatory disease of the colon or rectum, or of unresolved occlusion or sub-occlusion for which symptomatic treatment is being administered
* Other concomitant cancer or history of cancer during the 5 years, with the exception of a carcinoma in situ of the cervix or basal cell or squamous cell carcinoma, considered cured
* Significant history of heart or respiratory disease, including any history of interstitial pneumonia
* Patient already included in another clinical trial with an experimental molecule
* Women who are breast-feeding
* Persons deprived of liberty or under guardianship
* Unable to submit to medical monitoring during the trial due to geographical, social or psychological reasons

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2021-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julien TAIEB, Pr, Study Chair — HEGP - PARIS - FRANCE
Locations (37):
- France (37):
  - Clinique Privée Claude Bernard, Albi
  - CH, Blois
  - Clinique Tivoli Ducos, Bordeaux
  - Hôpital Duchenne, Boulogne-sur-Mer
  - CH Pierre Oudot, Bourgoin
  - Centre François Baclesse, Caen
  - CHR côte de Nacre, Caen
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Centre GF Leclerc, Dijon
  - CH de la Dracénie, Draguignan
  - Ch Jacques Monod, Flers
  - CH, Fréjus
  - CHU, Le Kremlin-Bicêtre
  - CH, Le Mans
  - CHU, Limoges
  - Clinique Chenieux, Limoges
  - CH, Longjumeau
  - CH Pierre Benite, Lyon
  - Hopital Europeen Marseille, Marseille
  - H Layné, Mont-de-Marsan
  - HEGP, Paris
  - Hôpital La Pitié Salpêtrière, Paris
  - Hôpital Cochin, Paris
  - CH St Jean, Perpignan
  - Hôpital Haut Lévèque, Pessac
  - Centre Cario - Hpca Saint Brieuc, Plérin
  - Hôpitaux Drome Nord, Romans-sur-Isère
  - CHU, Rouen
  - CHP, Saint-Grégoire
  - Clinique Privée, Strasbourg
  - Hopitaux Du Leman, Thonon-les-Bains
  - Clinique Pasteur Groupe ONCORAD GARONNE, Toulouse
  - Clinique Privée Pasteur, Toulouse
  - Clinique Privée Saint Jean, Toulouse
  - Clinique St Jean Languedoc, Toulouse
  - Gustave Roussy, Villejuif
  - Hôpital Paul Brousse, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Rinaldi Y, Pointet AL, Khemissa Akouz F, Le Malicot K, Wahiba B, Louafi S, Gratet A, Miglianico L, Laharie H, Bouhier Leporrier K, Thirot Bidault A, Texereau P, Coriat R, Terrebonne E, Gouttebel MC, Malka D, Bachet JB, Lepage C, Taieb J; PRODIGE 37 Investigators/Collaborators. Gemcitabine plus nab-paclitaxel until progression or alternating with FOLFIRI.3, as first-line treatment for patients with metastatic pancreatic adenocarcinoma: The Federation Francophone de Cancerologie Digestive-PRODIGE 37 randomised phase II study (FIRGEMAX). Eur J Cancer. 2020 Sep;136:25-34. doi: 10.1016/j.ejca.2020.05.018. Epub 2020 Jul 2. PMID 32623182

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 2015 and November 2016, 127 patients were enrolled in the trial by 36 french centres .
Groups:
- Nab-paclitaxel + Gemcitabine/FOLFIRI.3: Alternance of :
  * 2 months with nab-paclitaxel (125 g/m² - 30 min in IV) + gemcitabine (1000 mg/m², 30 min in IV, 3 injections follow by 1 week free)
  * follow by 2 months with FOLFIRI.3 (irinotecan: 90 mg/m² at D1, acid folinic 400 mg/m², 5Fu continus: 2000 mg/m² IV 46 hours, and irinotecan at D3, 90 mg/m²) This alternance continus until progression
  FOLFIRI.3: For each cycle : 1 week out of 2 - injection at Day1, J15 Irinotécan 90 mg/m² at day1 in perfusion over 60 min in Y of folinic acid Folinic Acid 400 mg/m² (or 200 mg/m² Elvorine) at Day 1 in perfusion over 2 hours 5FU continu 2000 mg/m² during 46 hours Irinotécan at 90 mg/m² in perfusion over 60 mn at Day 3 (when 5FU perfusion is over)
  nab-paclitaxel+ gemcitabine: For each cycle : 3 weeks out of 4 - injection at Day 1, 8 and 15 Nab-paclitaxel : 125 mg/m² of nab-paclitaxel in perfusion over 30 mn. Gemcitabine 1000 mg/m² in perfusion over 30 mn immediately after Nab paclitaxel administration is over.
Period: Overall Study
Arm/Group | Nab-paclitaxel + Gemcitabine/FOLFIRI.3 | Nab-paclitaxel + Gemcitabine
Started | 64 | 63
Completed | 62 | 60
Not Completed | 2 | 3
Not completed — Death | 1 | 2
Not completed — Patients not treated | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline description is done on the ITT population meaning all the randomized patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nab-paclitaxel + Gemcitabine/FOLFIRI.3 | Nab-paclitaxel + Gemcitabine | Total
Number analyzed (Participants) | 64 | 63 | 127
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 34 | 33 | 67
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65.20 [57.66 to 69.70] | 65.99 [59.42 to 69.54] | 65.33 [58.89 to 69.54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 34 | 62
  Male | 36 | 29 | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 64 | 63 | 127
Region of Enrollment [Number; unit: participants]
  France | 64 | 63 | 127

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Alive and Without Radiological and/or Clinical Progression 6 Months After the Randomization
Description: The primary endpoint was the rate of patients alive and progression-free 6 months after randomization.
  Progression was assessed by the investigator and defined radiologically according to RECIST v1.1 criteria and/or clinically as deterioration of general condition not related to treatment, palpable tumor masses on clinical examination (adenopathy, tumor hepatomegaly, peritoneal carcinosis), pleural effusion, ascites.
  Patients who progressed or died before 6 months were considered to have failed the primary endpoint at 6 months.
  The 6-month imaging was the imaging done at 6 months with a +/- 1 month window.
Time Frame: 6 months after randomization
Population: The primary endpoint was analysed on the mITT population meaning all the randomized patients with at least one dose of study drug taken
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-paclitaxel + Gemcitabine/FOLFIRI.3 | Nab-paclitaxel + Gemcitabine
Number analyzed (Participants) | 62 | 60
Participants | 28 | 14

2. Secondary Outcome: Overall Survival (OS):
Description: Overall survival was defined as the time from the date of randomization to the patient's death (all causes). For alive patients, the date of last news was taken into account
Time Frame: Up to 2 years after the treatment start
Population: Endpoint was analyzed on the ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-paclitaxel + Gemcitabine/FOLFIRI.3 | Nab-paclitaxel + Gemcitabine
Number analyzed (Participants) | 64 | 63
months | 11.71 [7.92 to 14.55] | 10.94 [8.18 to 12.39]

3. Secondary Outcome: Best Response
Description: Best response is defined as the best response for each patient regarding imagerie taken during the treatment. Response was evalauted according to RECIST v1.1 over the entire treatment period according the investigator
Time Frame: Up to the end of treatment on the average of 12 months
Population: Endpoint was analysed on mITT population meaning all randomized patients having at least one dose of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-paclitaxel + Gemcitabine/FOLFIRI.3 | Nab-paclitaxel + Gemcitabine
Number analyzed (Participants) | 62 | 60
Participants
  Complete response | 1 | 0
  Partial Response | 24 | 16
  Stability | 20 | 26
  Progression | 5 | 13
  Death without any imagery | 12 | 5

4. Secondary Outcome: Progression-free Survival (PFS)
Description: It was defined as the time between t randomization and the date of the first radiological progression (RECIST 1.1 criteria) and/or clinical progression according to the investigator or death (whatever the cause is); Patients alive without progression were censored at date of last news
Time Frame: up to 12 months after randomization
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-paclitaxel + Gemcitabine/FOLFIRI.3 | Nab-paclitaxel + Gemcitabine
Number analyzed (Participants) | 64 | 63
months | 5.72 [3.68 to 7.59] | 4.21 [2.43 to 6.01]

ADVERSE EVENTS:
Time Frame: Both deaths and adverse events were assessed up to 2 years
Description: Adverse events were analyzed on the population of patients who received at leats one dose of treatment and regarding the treatment really received by the patient. Two patients randomized in the Nab-paclitaxel + Gemcitabine arm received Nab-paclitaxel + Gemcitabine - Folfiri. So, these patient wereanalyzed in the Nab-paclitaxel + Gemcitabine/FOLFIRI.3 arm for tolerance
  For all cause of mortality, the population was the ITT population meaning all patients randomized.
Arm/Group | Nab-paclitaxel + Gemcitabine/FOLFIRI.3 | Nab-paclitaxel + Gemcitabine
All-Cause Mortality (participants affected / at risk) | 53/64 | 54/63
Serious Adverse Events (participants affected / at risk) | 30/64 | 19/58
Other Adverse Events (participants affected / at risk) | 63/64 | 58/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nab-paclitaxel + Gemcitabine/FOLFIRI.3 (N=64) | Nab-paclitaxel + Gemcitabine (N=58)
Cardiac arrest (Cardiac disorders) | 0 | 2
Transient Ischemic Attack (Nervous system disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 1
Hypocellular bone marrow (Blood and lymphatic system disorders) | 2 | 1
Venous thromboembolic event (Vascular disorders) | 1 | 2
Thromboembolic event (Vascular disorders) | 1 | 1
Catheter infection (Infections and infestations) | 4 | 2
Biliary tract infection (Hepatobiliary disorders) | 2 | 2
Septicemia (Infections and infestations) | 5 | 6
Hypokaliemia (Metabolism and nutrition disorders) | 3 | 0
Multivisceral failure (General disorders) | 1 | 0
Fatigue (General disorders) | 5 | 5
Thrills (General disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nab-paclitaxel + Gemcitabine/FOLFIRI.3 (N=64) | Nab-paclitaxel + Gemcitabine (N=58)
Vertigo (Ear and labyrinth disorders) | 5 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 31 | 32
Palmo-palmar syndrome (Skin and subcutaneous tissue disorders) | 8 | 3
Allergic reaction (Immune system disorders) | 6 | 4
Cephalgia (Nervous system disorders) | 4 | 7
Paresthesia (Nervous system disorders) | 22 | 23
Dysgueusia (Nervous system disorders) | 5 | 5
Constipation (Gastrointestinal disorders) | 15 | 18
Diarrhea (Gastrointestinal disorders) | 45 | 35
Mucitis (Gastrointestinal disorders) | 14 | 12
Nausea (Gastrointestinal disorders) | 42 | 30
Vomiting (Gastrointestinal disorders) | 30 | 21
Abdominal pain (Gastrointestinal disorders) | 25 | 16
Anemia (Blood and lymphatic system disorders) | 58 | 55
Sensitive neuropathie peripheral (Nervous system disorders) | 15 | 16
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Venous thromboembolic event (Vascular disorders) | 10 | 6
Anorexia (Metabolism and nutrition disorders) | 38 | 26
Fatigue (General disorders) | 57 | 49
Fever (General disorders) | 24 | 18
Inferior members oedema (General disorders) | 16 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-12-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT02827201/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT02827201/SAP_001.pdf